CLINICAL TRIAL: NCT05927441
Title: Safety and Performance Evaluation Study of DragonFly System for Mitral Regurgitation
Brief Title: DragonFly EU Pivotal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Collaborators: Donawa Lifescience (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DJ/TD/08CC-01E
Record Dates: First submitted 2023-06-17; First posted 2023-07-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DragonFly Transcatheter Mitral Valve Repair System-DMR (Experimental): Transcatheter mitral valve repair with the DragonFly System in patients with degenerative mitral regurgitation
  Interventions: Device: DragonFly Transcatheter Mitral Valve Repair System
- DragonFly Transcatheter Mitral Valve Repair System-FMR (Experimental): Transcatheter mitral valve repair with the DragonFly System in patients with functional mitral regurgitation
  Interventions: Device: DragonFly Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: DragonFly Transcatheter Mitral Valve Repair System — Edge-to-edge repair with DragonFly System
  Other Names: Transcatheter Mitral Valve repair (TMVr)

SUMMARY:
To confirm the effectiveness and safety of the DragonFly Transcatheter Mitral Valve Repair System for the treatment of symptomatic moderate-to-severe (3+) or severe (4+) degenerative mitral regurgitation in high surgical risk subjects and symptomatic moderate-to- severe (3+) or severe (4+) functional mitral regurgitation subjects who remained clinically symptomatic after adequate treatment.

DETAILED DESCRIPTION:
This is a prospective, multicentric clinical investigation.

Subjects to be included in this clinical investigation suffer from symptomatic chronic moderate-to-severe (3+) or severe (4+) DMR with high or prohibitive surgical risk judged by a local investigation site's heart team and symptomatic moderate-to- severe (3+) or severe (4+) functional mitral regurgitation subjects who remained clinically symptomatic after adequate treatment.

Local heart teams must include at a minimum a cardiac surgeon experienced in mitral valve surgery and a cardiologist experienced in mitral valve disease. After signing the informed consent form (ICF), a subject will be enrolled and treated with the DragonFlyTM Transcatheter Mitral Valve Repair System (Valgen Medtech, Hangzhou).

The CE-DMR cohort clinical investigation will be assessed at the following intervals: implant, before discharge, 30 days, 6 months and annually for 5 years. Group sequential design analysis is planned based on an adaptive design to assess whether the primary endpoint will be met. If the primary endpoint is not met at the interim analysis, then it will be re-analyzed for 160 patients when all subjects in Europe/Canada complete 12 months follow-up.

The CE-FMR cohort clinical investigation will be assessed at the following intervals: implant, before discharge, 30 days, 6 months and annually for 5 years. An adaptive design with sample size re-estimation will be incorporated. The primary endpoint will be assessed at the interim analysis. If the conditional power falls within the promising zone (38-80%), then the sample size will be re-estimated to maintain at least 80% power. Then the primary endpoint will be evaluated once the 12-month follow-up is completed with the larger sample size (not less than 165).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* New York Heart Association (NYHA) Class II-IV
* Moderate to severe (3+) or severe (4+) chronic DMR determined by transthoracic echocardiography (For DMR cohort)
* Symptomatic FMR ≥ 3+ due to ischemic or non-ischemic cardiomyopathy (For FMR cohort)
* Transseptal catheterization and femoral vein access are determined to be feasible
* Subjects have been informed of the nature of the study, understand the purpose of the clinical trial, voluntarily participate in the study, and sign the ICF

Exclusion Criteria:

* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Other severe heart valve diseases requiring intervention
* Prior mitral valve leaflet surgery (prior annuloplasty ring not excluded) or previous transcatheter mitral valve intervention
* Acute myocardial infarction occurred within 4 weeks, or untreated severe coronary artery stenosis requiring revascularization
* Any cardiovascular intervention within 30 days or cardiac surgery within 6 months prior to the procedure; or in the judgment of the investigator, the femoral vein cannot accommodate a 25 F catheter or the presence of an inferior vena cava filter would interfere with advancement of the catheter or ipsilateral deep vein thrombosis is present; or the patient's anatomy is not suitable for atrial septal puncture
* Patients in whom TEE or general anesthesia is contraindicated
* End stage heart failure (ACC/AHA stage D); or after heart transplantation; or waiting for a heart transplantation
* Active endocarditis or active rheumatic heart disease; or mitral valve changes due to endocarditis and rheumatic heart valve disease
* History of ischemia cerebrovascular accident in the past 30 days, or severe symptomatic carotid stenosis (ultrasonic examination showed stenosis degree >70%); or carotid stent implantation within 30 days; hemorrhagic cerebrovascular accident occurred within 6 months
* History of acute peptic ulcer or gastrointestinal bleeding within 3 months
* Hemorrhagic disease or coagulation disorder; or contraindicated of antithrombotic drug treatment
* Modified Rankin scale ≥ 4
* Diseases that make the evaluation of treatment difficult (e.g., cancer, severe metabolic disease, psychosis)
* Pregnant or lactating women
* Hemodynamic instability defined as systolic pressure < 90 mmHg without afterload reduction medicine, or cardiogenic shock, or need for an intra-aortic balloon pump, or other hemodynamic support devices
* Active infections requiring current antibiotic therapy (if temporary illness, patients may be enrolled 2 weeks after discontinuation of antibiotics)
* Currently participating in an investigational drug or another device study of which the primary endpoint has not been completed, or it that clinically interferes with the current study endpoints. (Note: extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational study)
* In the judgment of the investigator, the patients' compliance will be poor and could not complete the study as required, or other conditions indicate that the subject is not suitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 12 months after the procedure for DMR Cohort only | 12 months
  The rate of the composite endpoint of freedom from all-cause mortality, surgery for mitral valve dysfunction, or MR > 2+ at 12 months.
Freedom from all-cause mortality, or hospitalization for heart failure events at 12 months after the procedure for FMR Cohort only | 12 months
  Freedom from all-cause mortality, or hospitalization for heart failure events at 12 months after the procedure for FMR Cohort only

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maisano, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Universitatsklinikum Bonn Medizinische Klinik und Poliklinik, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No